CLINICAL TRIAL: NCT04661462
Title: Health After COVID-19 in the European Region Tyrol - South Tyrol
Brief Title: Health After Covid-19 in Tyrol
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Collaborators: Claudiana Landesfachhochschule (Other)
Responsible Party: Sponsor
Other Study IDs: 20200928-2379
Record Dates: First submitted 2020-09-29; First posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-09

CONDITIONS: COVID-19
Keywords: long term sequelae
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

INTERVENTIONS:
Other: online survey — We invite volunteers after COVID-19 to participate in an online survey.

SUMMARY:
The aim of the regional online questionnaire is to better understand the pattern of acute infection and the time of recovery of various symptoms.

DETAILED DESCRIPTION:
The ongoing COVID-19 pandemic considerably increases the demand for healthcare and raises concerns on longterm disease outcome. Accordingly, to increase the knowledge on recovery from symptoms of acute infection and longterm health effects, a regional COVID-19 online survey on the health-status after infection will be performed.

This cross-sectional anonymous online survey is initiated and conducted by an interdisciplinary study team of the Medical University of Innsbruck, Austria.

For each participant, demographic characteristics (e.g. age, gender, district affiliation, profession), medical history (presence of comorbidities, medication), diagnosis of COVID-19, symptoms and their duration, treatments and special conditions will be collected.

The aim of the survey is to better understand the pattern of acute infection and the time of recovery of various symptoms.

The anonymous online survey is open to individuals after COVID-19 infection (proven by SARS-Cov-2 positive PCR or antibody test) over the age of 16 and living in Tyrol (Western-Austria).

The survey takes around 30 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* status post COVID-19 infection, defined by a positive SARS-Cov-2 PCR or antibody test
* age ≥ 16years
* resident in Tyrol (Austria)

Exclusion Criteria:

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: voluntary participation of probands after COVID-19, resident in Tyrol, Austria, with access to online survey;
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Population based data on spectrum and recovery from COVID-19 symptoms | two weeks after infection
  Percentage of patients manifesting ongoing symptoms after 2 weeks of infection.
Population based data on spectrum and recovery from COVID-19 symptoms | up to 24 weeks
  Spectrum of symptoms at onset and at end of disease.
Predictors of recovery. | up to 24 weeks
  Identification of symptoms or comorbidities associated with Long-Covid-19.

CONTACTS AND LOCATIONS:
Locations (1):
- Medizinische Universität Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rass V, Tymoszuk P, Sahanic S, Heim B, Ausserhofer D, Lindner A, Kofler M, Mahlknecht P, Boehm A, Hufner K, Pizzini A, Sonnweber T, Kurz K, Pfeifer B, Kiechl S, Peball M, Kindl P, Putnina L, Fava E, Djamshidian A, Huber A, Wiedermann CJ, Sperner-Unterweger B, Woll E, Beer R, Schiefecker AJ, Bellmann-Weiler R, Bachler H, Tancevski I, Pfausler B, Piccoliori G, Seppi K, Weiss G, Loffler-Ragg J, Helbok R. Distinct smell and taste disorder phenotype of post-acute COVID-19 sequelae. Eur Arch Otorhinolaryngol. 2023 Nov;280(11):5115-5128. doi: 10.1007/s00405-023-08163-x. Epub 2023 Sep 5. PMID 37670171
- [Derived] Hufner K, Tymoszuk P, Ausserhofer D, Sahanic S, Pizzini A, Rass V, Galffy M, Bohm A, Kurz K, Sonnweber T, Tancevski I, Kiechl S, Huber A, Plagg B, Wiedermann CJ, Bellmann-Weiler R, Bachler H, Weiss G, Piccoliori G, Helbok R, Loeffler-Ragg J, Sperner-Unterweger B. Who Is at Risk of Poor Mental Health Following Coronavirus Disease-19 Outpatient Management? Front Med (Lausanne). 2022 Mar 14;9:792881. doi: 10.3389/fmed.2022.792881. eCollection 2022. PMID 35360744